CLINICAL TRIAL: NCT04719507
Title: Ultrasound Guided Erector Spinae Block Versus Thoracic Paravertebral Block for Postoperative Pain Control After Open Nephrectomy : A Randomized Controlled Trial
Brief Title: Erector Spinae Block Versus Thoracic Paravertebral Block for Postoperative Pain Control After Open Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ezzat Ramzy Ezz, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: pain control in nephrectomy
Record Dates: First submitted 2021-01-09; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
Keywords: open nephrectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- erector spinae arm (Experimental): ultrasound guided erector spinae block
  Interventions: Procedure: erector spinae block
- thoracic paravertebral arm (Experimental): ultrasound guided thoracic paravertebral block.
  Interventions: Procedure: thoracic paravertebral block
- drug arm (Active Comparator): pethidine (1 mg/kg ) once
  Interventions: Drug: Pethidine Only Product in Parenteral Dose Form

INTERVENTIONS:
Procedure: erector spinae block — ultrasound probe is placed parallel to the vertebral spine at T4 level and shifted 3 cm laterally to obtain the appropriate visualization. Under aseptic precautions, the needle is inserted and advanced perpendicular to the skin in all planes to contact the transverse process of the vertebra at a variable depth of 2-4 cm from the skin depending on the build of the individual. At this point, the needle tip lies between the erector spinae muscle and transverse process. After negative aspiration, 20 ml of 0.25% bupivacaine is administered in cephalad and caudal directions.
  Other Names: erector spinae plane block
  Arms: erector spinae arm
Procedure: thoracic paravertebral block — ultrasound probe is placed parallel to the vertebral spine at T4 level and shifted 2-3 cm laterally to obtain the appropriate visualization. Following the identification of pleura, transverse process and paravertebral space, the needle is inserted cranial to caudal direction using in-plane approach . After confirming the displacement of pleura with 0.5-1 ml of local anesthetic (LA), 20 ml of 0.25% bupivacaine is administered for the block.
  Arms: thoracic paravertebral arm
Drug: Pethidine Only Product in Parenteral Dose Form — pethidine (1 mg/kg ) once
  Arms: drug arm

SUMMARY:
the study aims to compare the analgesic efficacy of erector spinae plane block versus thoracic paravertebral block after open nephrectomy surgery.

DETAILED DESCRIPTION:
Open nephrectomy is associated with substantial postoperative pain, pain relief in patients undergoing this procedure is usually provided either by thoracic epidural analgesia (EA) or systemic analgesics. EA is a very useful option for the management of postoperative pain in patients undergoing abdominal surgeries, but the risks and contraindications linked to EA like hypotension ,headache ,nerve damage or infection may limit its use. Systemic analgesics in the form of opioid analgesics may give rise to side effects like nausea ,vomiting ,constipation, allergy or drowsiness and often provide insufficient analgesia. Hence, other methods of postoperative pain management are desired. Sensory level target according to the incision site Flank(T9-T11) , Thoraco-abdominal (T7-T12 ) and Trans-abdominal (T6-T10).

Ultrasound (US) guided erector spinae plane (ESP) block is one of the interfascial plane blocks that target the dorsal and ventral rami of the spinal nerves. Although there is no sufficient evidence for the spread of local anesthetic to the ventral rami, recent anecdotal reports demonstrated effective postoperative analgesia after thoracic and lumbar surgeries affecting both the ventral and dorsal rami .According to a previous study, Erector Spinae Plane block has allowed a reduction in opioid consumption and excellent pain control in partial nephrectomy.

Paravertebral block (PVB) is a technique where a local anesthetic is deposited into a space found on both sides of the spine, called the paravertebral space. It is a block with a dermatomal distribution of pain relief depending on the level of the spine at which the block is sited and the quantity and type of deposited local anesthetic.

PVB is effective for pain relief in the thoracic, abdominal and limb regions .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (30-60 years) .
* Patients with ASA I , II score

Exclusion Criteria:

* Patient's refusal
* Coagulopathy to be cancelled if ( INR>1.4 , Platelets count <100x109 )
* Infection at the injection site.
* Allergy to local anesthetics.
* Patients receiving opioids for chronic analgesic therapy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Total morphine requirements 24 hours postoperatively | 24 hours postoperative
  morphine increment ( 0.02 mg/kg IV ) will be added to maintain a resting visual analogue score at <3 and the total 24-hours morphine consumption will be recorded

SECONDARY OUTCOMES:
Visual analogue score at 2, 4, 6, 12, 18, and 24 hours postoperatively | 2, 4, 6, 12, 18, and 24 hours postoperatively
  the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity .no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Time span to the first postoperative analgesia | calculated from the time of intervention till the time of the first rescue dose of morphine,expected form 2-3 hours
  Time span to the first postoperative analgesic request to be started from the time of the block till the first rescue dose of morphine
operation time | from start of anesthesia till the end of surgery , expected from 3-4 hours
  Duration of the anesthesia and surgery to be documented

REFERENCES:
- [Background] Gautam SKS, Das PK, Agarwal A, Kumar S, Dhiraaj S, Keshari A, Patro A. Comparative Evaluation of Continuous Thoracic Paravertebral Block and Thoracic Epidural Analgesia Techniques for Post-operative Pain Relief in Patients Undergoing Open Nephrectomy: A Prospective, Randomized, Single-blind Study. Anesth Essays Res. 2017 Apr-Jun;11(2):359-364. doi: 10.4103/0259-1162.194559. PMID 28663622
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698
- [Background] Kehlet H, Rung GW, Callesen T. Postoperative opioid analgesia: time for a reconsideration? J Clin Anesth. 1996 Sep;8(6):441-5. doi: 10.1016/0952-8180(96)00131-6. PMID 8872683
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Bonvicini D, Tagliapietra L, Giacomazzi A, Pizzirani E. Bilateral ultrasound-guided erector spinae plane blocks in breast cancer and reconstruction surgery. J Clin Anesth. 2018 Feb;44:3-4. doi: 10.1016/j.jclinane.2017.10.006. Epub 2017 Oct 21. No abstract available. PMID 29065335
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Santonastaso DP, de Chiara A, Musetti G, Bagaphou CT, Gamberini E, Agnoletti V. Ultrasound guided erector spinae plane block for open partial nephrectomy: only an alternative? J Clin Anesth. 2019 Sep;56:55-56. doi: 10.1016/j.jclinane.2019.01.036. Epub 2019 Jan 25. No abstract available. PMID 30690313
- [Background] Karmakar MK, Samy W, Lee A, Li JW, Chan WC, Chen PP, Tsui BCH. Survival Analysis of Patients with Breast Cancer Undergoing a Modified Radical Mastectomy With or Without a Thoracic Paravertebral Block: a 5-Year Follow-up of a Randomized Controlled Trial. Anticancer Res. 2017 Oct;37(10):5813-5820. doi: 10.21873/anticanres.12024. PMID 28982906
- [Background] Chu L, Zhang X, Lu Y, Xie G, Song S, Fang X, Cheng B. Improved Analgesic Effect of Paravertebral Blocks before and after Video-Assisted Thoracic Surgery: A Prospective, Double-Blinded, Randomized Controlled Trial. Pain Res Manag. 2019 Nov 18;2019:9158653. doi: 10.1155/2019/9158653. eCollection 2019. PMID 31827657
- [Background] Greengrass R, Buckenmaier CC 3rd. Paravertebral anaesthesia/analgesia for ambulatory surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):271-83. doi: 10.1053/bean.2002.0238. PMID 12491557
- [Background] Baik JS, Oh AY, Cho CW, Shin HJ, Han SH, Ryu JH. Thoracic paravertebral block for nephrectomy: a randomized, controlled, observer-blinded study. Pain Med. 2014 May;15(5):850-6. doi: 10.1111/pme.12320. Epub 2013 Dec 16. PMID 24341324
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Forastiere E, Sofra M, Giannarelli D, Fabrizi L, Simone G. Effectiveness of continuous wound infusion of 0.5% ropivacaine by On-Q pain relief system for postoperative pain management after open nephrectomy. Br J Anaesth. 2008 Dec;101(6):841-7. doi: 10.1093/bja/aen309. PMID 19004914